CLINICAL TRIAL: NCT04309851
Title: A Deep Learning Approach to Submerged Deciduous Teeth Classification and Detection
Brief Title: A Deep Learning Approach to Submerged Teeth Classification and Detection
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Seçil Çalışkan, Assistant Professor, Eskisehir Osmangazi University
Other Study IDs: E86412-49
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Artificial Intelligence; Submerging Tooth
Keywords: artificial intelligence; infraocclusion; submerged tooth
MeSH Terms: interventions — Deep Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: deep learning — the deep learning method is a field of study involving artificial neural networks and similar machine learning algorithms with many hidden layers.

SUMMARY:
Objectives: The study aimed to compare the success and reliability of an artificial intelligence application in the detection and classification of submerged teeth in orthopantomography (OPG).

Methods: Convolutional neural networks (CNN) algorithms were used to detect and classify submerged molars. The detection module, which is based on the state-of-the-art Faster R-CNN architecture, processed the radiograph to define the boundaries of submerged molars. A separate testing set was used to evaluate the diagnostic performance of the system and compare it to the expert level.

Results: The success rate of classification and identification of the system is high when evaluated according to the reference standard. The system was extremely accurate in performance comparison with observers.

Conclusions: The performance of the proposed computer-aided diagnosis solution is comparable to that of experts. It is useful to diagnose submerged molars with an artificial intelligence application to prevent errors. Also, it will facilitate pediatric dentists' diagnoses.

DETAILED DESCRIPTION:
Pre-processing, Training, and Classification The study was conducted with balanced data sets. The case and control data sets were randomly divided into two parts, the training group (27 case group/27 control group) and the test group (10 case group/10 control group) to prevent the use of the visuals in the training group for retesting. The testing data set was not seen by the system during the training phase.

All 2943-by-1435 pixel images in the data set were resized to 971 by 474 pixels prior to training. All OPG images used include the whole dentitions. The training and test data sets were used to estimate and generate weight factors for the optimal CNN algorithm. An arbitrary sequence was generated using open-source Python programming (Python 3.6.1, Python Software Foundation, Wilmington, DE, USA, https://www.python.org/) language and OpenCV, NumPy, Pandas, and Matplotlib libraries. In this study, Tensorflow for model development was used to classify submerged primary molars. InceptionV3 architecture was used as transfer learning, and the transfer values were saved in the cache. Then, fully connected layer and softmax classifiers were combined to form the final model layers. The training was carried out using 7000 steps with 16G RAM and a PC equipped with NVIDIA GeForce GTX 1050.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

OPG images of poor quality (metal artifact, artifacts due to position errors during shooting, etc.) were excluded.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The data set included OPGs of 19000 children aged 5-12 years that were collected between January 2016 and December 2018.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Submerged Tooth Detection | 6 months
  The detection module, which is based on the state-of-the-art Faster R-CNN architecture, processed the radiograph to define the boundaries of submerged molars.

CONTACTS AND LOCATIONS:
Locations (1):
- Seçil Çalışkan, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided